CLINICAL TRIAL: NCT06408454
Title: Determination of IL-17, Bcl-3, AND IκBζ Expression Levels in the Gingival Crevicular Fluid of Psoriasis Patients
Brief Title: Interleukin- 17 (IL-17), Bcl-3, and NF-kappa-B Inhibitor Zeta (IκBζ) Expression Levels in the Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, AYŞE GÜL ÖNER TALMAÇ, assistant professor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU-ONERTALMAC-01
Record Dates: First submitted 2024-04-15; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis; Periodontal Diseases
Keywords: psoriasis; gene expression; periodontal health
MeSH Terms: conditions — Psoriasis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriasis patients: IL-17, Bcl-3, IκBζ gene expression levels were examined
  Interventions: Diagnostic Test: Gingival crevicular fluid collection; Diagnostic Test: periodontal test
- Control group: IL-17, Bcl-3, IκBζ gene expression levels were examined
  Interventions: Diagnostic Test: Gingival crevicular fluid collection; Diagnostic Test: periodontal test

INTERVENTIONS:
Diagnostic Test: Gingival crevicular fluid collection — Samples were taken from two mandibular molar teeth. Before sampling, the sites were isolated with cotton rolls and then carefully dried with an air syringe to avoid saliva contamination. GCF was collected using sterile periodontal strips by gently inserting them into the gingival sulcus or pocket until slight resistance was noticed. After 30 s, the strips were collected into sterile tubes and immediately transported to the laboratory for storage (-40 °C) and posterior analysis.
Diagnostic Test: periodontal test — A periodontist conducted the periodontal evaluation, which included a comprehensive assessment of clinical periodontal status, a full mouth manual periodontal charting, measurement of probing depth, clinical attachment level, bleeding on probing, and evaluation of mobility using a periotest device. Additionally, information regarding the patient's smoking status, frequency of smoking, and oral hygiene habits was obtained.

SUMMARY:
This study aimed to compare the levels of IL-17 (interleukin- 17), Bcl-3 (B-cell lymphoma 3-encoded protein), and IκBζ (NF-kappa-B inhibitor zeta) in the gingival crevicular fluid of psoriatic and healthy individuals and the clinical parameters such as periodontal health, gingival index, plaque index and mobility (using periotest device)in the patient and control groups.

DETAILED DESCRIPTION:
Patient selection

Ten patients previously diagnosed with psoriasis who visited the Van 100. Yıl University Faculty of Dentistry Oral and Maxillofacial Radiology dental clinic were included in the study. Non-psoriasis individuals were selected from volunteer patients attending the same dental clinic.

Clinical measurements

A periodontist conducted the periodontal evaluation, which included a comprehensive assessment of clinical periodontal status, a full mouth manual periodontal charting, measurement of probing depth, clinical attachment level, bleeding on probing, and evaluation of mobility using a periotest device. Additionally, information regarding the patient's smoking status, frequency of smoking, and oral hygiene habits was obtained.

Gingival crevicular fluid (GCF) collection

Samples were taken from two mandibular molar teeth. Before sampling, the sites were isolated with cotton rolls and then carefully dried with an air syringe to avoid saliva contamination. GCF was collected using sterile periodontal strips by gently inserting them into the gingival sulcus or pocket until slight resistance was noticed. After 30 s, the strips were collected into sterile tubes and immediately transported to the laboratory for storage (-40 °C) and posterior analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with psoriasis
* Adults who are 18 years of age or older
* Patients having at least 11 teeth

Exclusion Criteria:

* Patients with any known systemic disease other than psoriasis
* Patients who had received antibiotic, nonsteroidal anti-inflammatory, and/or immunomodulatory therapy within the last three months
* Patients who had received radiotherapy and/or chemotherapy within the last years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients living in Eastern region of Turkey and visiting our clinic
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Level of Gene expression | Sample collection during examination, approximately 2 months
  In the real-time polymerase chain reaction (PCR) results of the β-actin gene, which was used as a housekeeping gene in the study, the automatic threshold value was determined by the device as 0.02. It was observed that all samples were above the threshold value and gave a ct value. According to the housekeeping gene, IL-17, IκBζ, and Bcl-3gene expression values were determined.

SECONDARY OUTCOMES:
Plaque index | Baseline, week 2
  To determine the plaque index of the patients, their dental plaque thickness was evaluated by probing surfaces of selected teeth using a periodontal probe. Scores range from 0 to 3.
Gingival index | Baseline, week 2
  To determine the gingival index of the patients, gingival bleeding caused by running a Williams periodontal probe inside the pocket on the mesial, distal, buccal, and palatal surfaces of selected teeth was evaluated. Scores range from 0 to 3.
Clinical attachment level | Baseline, week 2
  This parameter represents the extent of periodontal support that has been lost around a tooth and is measured with the periodontal probe as the distance from the cemento-enamel junction (CEJ) to the base of the pocket (in mm)
Tooth Mobility | Baseline, week 2
  The amount of tooth mobility can be displayed by a value called periotest value (PTV) ranging from -8 to +50

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Gül Öner Talmaç, PhD, Principal Investigator — Faculty of Dentistry, Kahraman Maraş Sütçü İmam University
Locations (1):
- Ayşe Gül Öner Talmaç, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No